CLINICAL TRIAL: NCT05146726
Title: Patient Blood Management Charité (PBM-Charité): ): Cohort Study About Structured Detection, Differentiated Diagnostics and Therapy of Preoperative Anemia and Use of Machine Autotransfusion in Elective Interventions
Brief Title: Patient Blood Management Charité (PBM-Charité): Structured Detection, Differentiated Diagnostics and Therapy of Preoperative Anemia and Use of Machine Autotransfusion in Elective Interventions
Status: Recruiting | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Claudia Spies, Head of the Department of Anesthesiology and operative Intensive Care (CCM/CVK), Charité- Universitätsmedizin Berlin, Charite University, Berlin, Germany
Other Study IDs: Patient Blood Management
Record Dates: First submitted 2021-11-16; First posted 2021-12-07 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-07

CONDITIONS: Anemia
Keywords: Transfusion; Machine autotransfusion
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prospective BARMER insured patients: Group I: BARMER insured patients with preoperative anemia and an elective (N5) surgical intervention with a probability of transfusion > 10%.
  Central measures in this group are the IV contract for the creation of an organizational and financing structure for the guideline-compliant detection, diagnosis and treatment of preoperative anemia and the evaluation of the machine autotransfusion as part of the preoperative premedication visit in anesthesiology (implementation is the responsibility of the patient blood management (PBM) service).
  Interventions: Other: BARMER anemia treatment
- Retrospective patients insured with another statutory health insurer than BARMER: Group II: Patients not insured with BARMER and with preoperative anemia and an elective (N5) surgical intervention with a probability of transfusion > 10% and receive early anemia detection.
  Interventions: Other: NON-BARMER anemia treatment

INTERVENTIONS:
Other: BARMER anemia treatment — BARMER insured patients are informed about the machine autotransfusion directly by the patient blood management (PBM) service and its intraoperative use is organized. The aim of these measures is to ensure that the intraoperative transfusion trigger does not fall below the intraoperative transfusion trigger by integrating the PBM into standard care and to avoid a perioperative transfusion. In addition, a postoperative treatment recommendation is made for the cause-related anemia treatment, e.g. in order to reduce the risk of a renewed anemia-related perioperative transfusion risk in the event of a possible follow-up operation or other elective operations.
  Groups: Prospective BARMER insured patients
Other: NON-BARMER anemia treatment — Patients not insured with BARMER also receive early anemia detection, selection according to indication intervention (transfusion probability> 10%) and evaluation for machine autotransfusion through the above-mentioned patient blood management (PBM) restructuring of standard care. In the case of preoperative anemia before an indication intervention and / or an intervention with machine autotransfusion application, the operating clinic will be given a recommendation by the PBM service for the diagnosis and treatment of the preoperative anemia and / or the use of the machine autotransfusion (implementation is the responsibility of the operating clinic)
  Groups: Retrospective patients insured with another statutory health insurer than BARMER

SUMMARY:
The aim of patient blood management is to reduce the risks of perioperative anemia- and transfusion-associated complications by limiting the use and the need for allogeneic blood transfusion.

DETAILED DESCRIPTION:
Background of this multimodal, multidisciplinary concept are numerous studies that have shown an association between preoperative anemia and/or a perioperative transfusion and a worse treatment outcome concerning morbidity and mortality. Diagnosis and therapy of preoperative anemia and the use of machine autotransfusion are central components of this integrated supply concept based on the S3 guideline "Präoperative Anämie", which need to be incorporated into the clinical processes.

Therefore, all patients undergoing elective surgery with a probability of transfusion > 10% receive an anemia detection during their premedication visit. Patients who are insured with BARMER also get anemia diagnostic and therapy. Patients of other health insurances receive a recommendation to anemia diagnostics and therapy sent to surgical department. Based on an analysis of the primary and secondary endpoints of this prospective cohort study, the implementation of the mentioned guideline-compliant measures in everyday clinical practice and the effectiveness of an IV-PBM (Patient blood management) are to be examined. Thus, if necessary, other health insurances could join the patient blood management (PBM) IV concept. The aim is to provide evidence of an improved quality of treatment and the generalized application of PBM measures within the scope of the innovative PBM care form described.

ELIGIBILITY:
Prospective:

Inclusion Criteria:

* age ≥ 18 years
* male and female patients
* patients eligible for inclusion: by the patient, preoperatively
* patients who are insured with BARMER
* patients with preoperative anemia and an elective (N5) surgical intervention with a probability of transfusion > 10%

additionally for the use of MAT:

* indication of machine autotransfusion
* high blood loss (> 500ml / 10-20 % of estimated blood volume) beside of indication interventions (surgery under dual platelet inhibition, high individual bleeding risk, special antibodies / rare blood group, rejection of allogeneic blood)

Exclusion Criteria:

* patients with emergency interventions
* rejection of study participation
* pregnancy, elective caesarean section or breastfeeding
* not enough German language skills
* accommodation in an institution because of judicial or administrative order
* employee of Charité
* missing of declaration of consent

Retrospective:

Inclusion Criteria:

-Data since September 2021-February 2024 of patients who are not insured with BARMER with elective (N5) interventions with a transfusion probability > 10% (indication list) with a preoperatively existing anemia

additionally for the use of MAT:

* indication of machine autotransfusion
* high blood loss (> 500ml / 10-20 % of estimated blood volume) beside of indication interventions (surgery under dual platelet inhibition, high individual bleeding risk, special antibodies / rare blood group, rejection of allogeneic blood)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with preoperative anemia and an electivesurgical intervention with a probability of transfusion > 10%
Sampling Method: Probability Sample
Enrollment: 2700 (Estimated)
Dates: Start 2022-02-02 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Number of patients | The participants are followed up until the end of hospital stay, an expected average of 7 days
  The amount of patients with differential diagnostics and causally appropriate therapy of a preoperative anemia of all patients with preoperative anemia before an elective surgical intervention with a probability of transfusion > 10% at study completion date = third year after start date (implementation rate of therapy recommendation). Approximately 9600 patients will be enrolled in the study. The data is evaluated after 3 years.

SECONDARY OUTCOMES:
Number of patients | The participants are followed up until the end of hospital stay, an expected average of 7 days
  The amount of patients with differential diagnostics and causally appropriate therapy of a preoperative anemia of all patients with preoperative anemia before an elective surgical intervention with a probability of transfusion > 10% after the first and second year after start date (implementation rate of therapy). The data of 2 is evaluated after 1 year and 2 years.
Number of machine autotransfusion respectively autologous transfusion | The participants are followed up until the end of hospital stay, an expected average of 7 days
  Number of patients which received machine autotransfusion
Rate of transfused patients | The participants are followed up until the end of hospital stay, an expected average of 7 days
  Number of patients which received transfusions
∆Hb before therapy of anemia and before surgical intervention | The participants are followed up until the end of hospital stay, an expected average of 7 days
  Difference between Hemoglobin before therapy of anemia and Hemoglobin before surgical intervention.
Number of allogeneic transfusions | The participants are followed up until the end of hospital stay, an expected average of 7 days
  Number of red cell concentrates per patient
Treatment period | The participants are followed up until the end of hospital stay, an expected average of 7 days
  Treatment period between begin of anemia therapy and surgical intervention
Treatment dose of anemia therapeutics in relation to ∆Hemoglobin | The participants are followed up until the end of hospital stay, an expected average of 7 days
  Treatment dose of anemia therapeutics in relation to the difference between Hemoglobin before begin of anemia therapy and the Hemoglobin before surgical intervention
Side effects 1 | The participants are followed up until the end of hospital stay, an expected average of 7 days
  Side effects of anemia therapeutics
Side effects 1 | The participants are followed up until the end of hospital stay, an expected average of 7 days
  Type of side effects of anemia therapeutics
Differences of secondary outcome measures | The participants are followed up until the end of hospital stay, an expected average of 7 days
  Differences of secondary outcome measures 2. - 10. mentioned above between long term and short term treatment (anemia therapy, long term treatment >3 weeks preoperative, short term treatment 1 - 3 days preoperative).
Anemia course | The participants are followed up until the end of hospital stay, an expected average of 7 days
  Change of Hemoglobin during hospital stay until hospital discharge
Length of hospital stay | The participants are followed up until the end of hospital stay, an expected average of 7 days
  Length of stay at the hospital
Length of intensive care unit stay | The participants are followed up until the end of hospital stay, an expected average of 3 days
  Length of stay at the intensive care unit
Rate and type of postoperative complications | The participants are followed up until the end of hospital stay, an expected average of 7 days
  Rate and type of Organ complications which are documented in the hospital records.
Side effects 2 | The participants are followed up until the end of hospital stay, an expected average of 7 days
  Type of side effects of machine autotransfusion
Rate of side effects | The participants are followed up until the end of hospital stay, an expected average of 7 days
  Rate of side effects of machine autotransfusion
Volumes of collected blood | The participants are followed up until the end of hospital stay, an expected average of 7 days
  Volumes of collected blood from Machine autotransfusion
Retransfused blood | The participants are followed up until the end of hospital stay, an expected average of 7 days
  Retransfused blood from Machine autotransfusion
Quality indicator 1 | The participants are followed up until the end of hospital stay, an expected average of 7 days
  Quality indicators for machine autotransfusion as process time
Quality indicator 2 | The participants are followed up until the end of hospital stay, an expected average of 7 days
  Quality indicators for machine autotransfusion as operating time
Quality indicator 3 | The participants are followed up until the end of hospital stay, an expected average of 7 days
  Quality indicators for machine autotransfusion as number of washing processes
Quality indicator 4 | The participants are followed up until the end of hospital stay, an expected average of 7 days
  Quality indicators for machine autotransfusion as surgery department
Quality indicator 5 | The participants are followed up until the end of hospital stay, an expected average of 7 days
  Quality indicators for machine autotransfusion as patient population
Rate of In-hospital mortality | The participants are followed up until the end of hospital stay, an expected average of 7 days
  Mortality is measured during hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Spies, MD, Prof., Study Director — Charite University, Berlin, Germany
Locations (1):
- Department of Anesthesiology and Operative Intensive Care Medicine (CCM/CVK), Charité - University Medicine Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No